CLINICAL TRIAL: NCT03033706
Title: Intraoperative Goal Directed Fluid Management Guided by Pulse Pressure Variation in Supratentorial Brain Tumor Craniotomy: a Randomized Controlled Study
Brief Title: Intraoperative Goal Directed Fluid Management in Supratentorial Brain Tumor Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Lecturer of anesthesia and critical care medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD-4-2016
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Brain Tumor; Craniotomy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Brain tumor excision under general anesthesia. Intervention (Pulse pressure variation guided fluid therapy): Study group will receive restricted fluid management with 1 ml/Kg/hr with concomitant PPV monitoring. PPV will be measured using invasive blood pressure monitor. Fluid bolus of 3 ml/Kg of ringer solution will be administrated whenever PPV is higher than 13%.
  Interventions: Procedure: Pulse pressure variation guided fluid therapy; Procedure: Brain tumor excision
- Control group (Placebo Comparator): Brain tumor excision under general anesthesia. Intervention (Traditional fluid therapy): Control Group will receive standard fluid management of 4 ml/Kg/hr ringer solution plus rescue fluid bolus of 200 ml Ringer solution if Mean arterial pressure decreased by 20% with central venous pressure less than 4 mmHg.
  Interventions: Procedure: Traditional fluid therapy; Procedure: Brain tumor excision

INTERVENTIONS:
Procedure: Pulse pressure variation guided fluid therapy — Pulse pressure variation obtained from invasive blood pressure waveform
  Arms: Study group
Procedure: Traditional fluid therapy — 4 ml/Kg/hr ringer solution plus rescue fluid bolus of 200 ml Ringer solution if Mean arterial pressure decreased by 20% with central venous pressure less than 4 mmHg.
  Arms: Control group
Procedure: Brain tumor excision — Brain tumor excision under general anesthesia

SUMMARY:
Pulse pressure variation (PPV) to standard fluid management (4ml/Kg/hr) in patients undergoing supratentorial mass excision. The investigators hypothesize that in these procedures, goal-directed fluid therapy (GDT) might improve brain relaxation, and patient hemodynamics intra and postoperatively.

DETAILED DESCRIPTION:
Neurosurgical operations are characterized by major fluid shift, frequent use of diuretics, and prolonged operative time. The role of fluid therapy in these patients is very critical, hypovolemia might lead to brain hypoperfusion and over-transfusion might lead increased intracranial tension. All these factors make fluid management in these procedures complex and challenging. Evidence on the optimum protocol for intraoperative fluid management in neurosurgical patients is still lacking.

Goal-directed therapy (GDT) in the operating room is a term used to describe the use of cardiac output or similar parameters to guide intravenous fluid and inotropic therapy.

Although GDT was well reported in many procedures, its benefit in neurosurgical operations is not well studied.

Pulse pressure variation (PPV) is a famous dynamic method of fluid responsiveness. PPV is simply calculated by dividing the largest pulse pressure (PPmax - PPmin) by the average pulse pressure (PPmax + PPmin /2) and expressed as percentage. PPV was previously used in GDT in major abdominal surgery with good performance.

The aim of this study is to compare the restricted fluid approach (1 ml/Kg/hr) guided by PPV to standard fluid management (4ml/Kg/hr) in patients undergoing supratentorial mass excision. The investigators hypothesize that in these procedures GDT might improve brain relaxation, and patient hemodynamics intra and postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for supratentorial mass excision will be enrolled in the study.

Exclusion Criteria:

* Patients with arrhythmias, pulmonary hypertension, impaired cardiac contractility, impaired liver or kidney function, and patients with BMI above 40 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of brain relaxation | one minute after dural puncture and one minute before dural closure
  A 4-point scale will be performed as follows: grade 1, perfectly relaxed; grade 2, satisfactorily relaxed; grade 3, firm brain; grade 4, bulging brain.

SECONDARY OUTCOMES:
volume of intraoperative fluid requirements | intraoperatively
  in litres
Urine output | intraoperatively
  Litres
heart rate | intraoperatively
  in beat per minute
number of episodes of hypotension | intraoperatively
  number of times where the blood pressure decreased by 25% of baseline
arterial blood gases | one hour postoperatively
  partial pressure of oxygen and carbon dioxide
serum lactate | one hour postoperatively
  in mmol per decilitre
Hemoglobin concentration | one hour postoperatively
  in grams per decilitre
prothrombin concentration | one hour postoperatively
  in percent

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No